CLINICAL TRIAL: NCT03642444
Title: Replacing Canes With an Elasticated Orthotic-garment in Chronic Stroke Patients: The Influence on Gait and Balance. A Series of N-of-1 Trials
Brief Title: Replacing Canes With an Elasticated Orthosis in Chronic Stroke Patients: The Influence on Gait and Balance. A Series of N-of-1 Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Bern (Other)
Collaborators: Bildungszentrum Gesundheit Basel-Stadt (Unknown); Rehab Basel (Other)
Responsible Party: Principal Investigator, Clare Maguire, Principle Investigator, Technical University of Bern
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TUBern
Record Dates: First submitted 2018-08-11; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: stroke; hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Canes

STUDY DESIGN:
Intervention Model Description: N-of-1 series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Phase A cane walking (assistive walking-device a cane) (Active Comparator): 9-12 weeks usual cane-walking to establish baseline values. Patients walk with their usual assistive-walking device - a cane.
  Interventions: Device: Cane
- Phase B elasticated orthotic-garment - TheraTogs (Active Comparator): 9-19 weeks : assistive walking-device which is an elasticated orthotic-garment worn throughout the day (product name TheraTogs). Cane use maximally reduced during his period.
  Interventions: Device: Elasticated worn orthotic-garment
- Phase C follow-Up (No Intervention): 9-10 weeks individually determined follow-up: subjects determine whether they walk independently (without assistive device) or with the elasticated orthotic-garment (TheraTogs) or with a cane.

INTERVENTIONS:
Device: Cane — Assistive walking device
  Arms: Phase A cane walking (assistive walking-device a cane)
Device: Elasticated worn orthotic-garment — Assistive walking device -elasticated worn orthotic garment
  Other Names: TheraTogs (product name)
  Arms: Phase B elasticated orthotic-garment - TheraTogs

SUMMARY:
This study aims to investigate the effect of an elasticated orthotic garment "Thera Togs" on walking ability and balance in currently cane using chronic stroke subjects (minimum 6 months post stroke) using a series of N-of-1 Trials.

DETAILED DESCRIPTION:
Aim: To investigate the effect of replacing canes with an elasticated orthotic-garment on gait and balance in chronic stroke subjects.

Design Experimental, multiple baseline N-of-1 series with an ABC design with randomised period duration.

Participants Four cane using chronic stroke subjects. Interventions Phase A (9-12 weeks) usual cane-walking to establish baseline values; Phase B (9-19 weeks) intervention: orthotic-garment worn throughout the day with maximal cane reduction; Phase C (9-10 weeks) individually determined follow-up: either no walking-aid, orthotic-garment or cane.

Weekly measurement of Outcome Measures for gait and balance function

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke (> six months since last stroke)
* Independent cane walkers. Subjects usually use canes to walk inside (this could be intermittent changing from cane to holding furniture etc.) and always when outside
* A Mini Mental Score of 22 or above.

Exclusion Criteria:

* Patients at risk of falling identified as a Berg Balance Score ≤42/56

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2014-10-15 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Functional Gait Assessment from baseline to post-Intervention (up to 28 weeks) | Post intervention up to 28 weeks (on average 21.5 weeks)
  Change of gait function between phases A (baseline) and Phase B (Intervention)

SECONDARY OUTCOMES:
Change in Trunk-sway from baseline to post-Intervention (up to 28 weeks) | Post intervention up to 28 weeks (on average 21.5 weeks)
  Change of trunk-sway at body center-of-mass during walking measured as Total-Angle-Area(TAA°) in frontal and sagittal-planes measured with a gyroscope "Sway Star" between phases A (baseline) and Phase B (Intervention)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maguire CC, Sieben JM, Lutz N, van der Wijden G, Scheidhauer H, de Bie R. Replacing canes with an elasticated orthotic-garment in chronic stroke patients - The influence on gait and balance. A series of N-of-1 trials. J Bodyw Mov Ther. 2020 Oct;24(4):203-214. doi: 10.1016/j.jbmt.2020.06.006. Epub 2020 Jul 30. PMID 33218513